CLINICAL TRIAL: NCT02122172
Title: Afatinib Dimaleate in Treating Patients With Advanced Refractory Urothelial Cancer
Brief Title: Afatinib in Advanced Refractory Urothelial Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to meet accrual goal after several years
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-0540; NCI-2014-00859 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB13-0540; 13-0540/ 1200.171 (Other: University of Chicago); P30CA014599 (NIH)
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Results first posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Distal Urethral Cancer; Proximal Urethral Cancer; Recurrent Bladder Cancer; Recurrent Urethral Cancer; Stage III Bladder Cancer; Stage III Urethral Cancer; Stage IV Bladder Cancer; Stage IV Urethral Cancer; Ureter Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms; Ureteral Neoplasms | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (afatinib) (Experimental): Patients receive afatinib dimaleate PO QD on days 1-42. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: afatinib dimaleate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: afatinib dimaleate — Given PO
  Other Names: afatinib; BIBW 2992 MA2; Gilotrif
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well afatinib dimaleate works in treating patients with urothelial cancer that cannot be removed surgically and has grown after treatment with standard first-line chemotherapy. Afatinib dimaleate may turn off the function of the epidermal growth factor (EGF) and human epidermal growth factor receptor 2 (HER2) receptors, which may slow the growth of cancer cells or cause some of the cells to die.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the 3-month progression free survival (PFS) rate in metastatic urothelial cancer patients receiving afatinib (afatinib dimaleate) who have progressed despite prior platinum-based chemotherapy.

SECONDARY OBJECTIVES:

I. To determine the overall response rate (complete response [CR] + partial response [PR]), median progression free survival, and overall survival for the same treated population.

II. To determine whether tumor epidermal growth factor receptor (EGFR) and/or HER2 overexpression influences 3-month PFS in patients treated with afatinib.

OUTLINE:

Patients receive afatinib dimaleate orally (PO) once daily (QD) on days 1-42. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have locally advanced or metastatic urothelial cancer that is not amenable to surgical treatment
* Patients must have histologically or cytologically confirmed urothelial tract carcinoma; patients with urothelial carcinoma of the bladder, upper tract, or urethra are eligible
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan for the evaluation of measurable disease (Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST v1.1])
* Patients must have evidence of disease progression prior to enrollment
* All patients must have received a prior platinum-based chemotherapy regimen for treatment of urothelial cancer and must now be considered refractory to platinum-based chemotherapy; patients may have received the platinum-containing regimen either in the peri-operative or metastatic setting
* Patients may have received up to one line of prior systemic chemotherapy for recurrent/metastatic disease; if a platinum-based regimen was received both in the peri-operative setting and again in the metastatic setting, this will be considered 1 line of chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 8.5g/dL
* Total bilirubin =< 1.5 institutional upper limit of normal (IULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X IULN
* Calculated creatinine clearance >= 30 mL/min by the modified Cockcroft and Gault Formula OR glomerular filtration rate >= 30 mL/min/body surface area (BSA) by Modification of Diet in Renal Disease or Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula
* Women and men of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients may not be receiving any other investigational agents
* Patients with untreated known brain metastases, or treated brain metastases that are clinically unstable
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements
* Women known to be pregnant
* Women who are breastfeeding and who are unwilling to stop breastfeeding prior to study entry
* Patients with known prior human immunodeficiency virus (HIV)-positive status on combination antiretroviral therapy are ineligible; known prior HIV-positive patients with CD4+ =< 500/mm^3 are ineligible (HIV testing is not required as part of this study)
* Pre-existing interstitial lung disease
* Inability to take oral medications
* Prior therapy with afatinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter O'Donnell, Principal Investigator — University of Chicago
Locations (6):
- United States (6):
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - NYU Langone Health, New York, New York
  - University of North Carolina - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Afatinib)
Started | 32
Main Phase II Study | 23
Molecularly Selected Cohort (Based on encouraging results from the main Phase II study, a molecularly selected cohort was enrolled) | 9
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Afatinib) - Phase II Study: Patients receive afatinib dimaleate PO QD on days 1-42. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
  afatinib dimaleate: Given PO
  Enrolled as part of the main Phase II study
- Treatment (Afatinib) - Molecularly Selected Cohort: Patients receive afatinib dimaleate PO QD on days 1-42. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
  afatinib dimaleate: Given PO
  Enrolled as part of the molecularly selected cohort
- Total: Total of all reporting groups
Arm/Group | Treatment (Afatinib) - Phase II Study | Treatment (Afatinib) - Molecularly Selected Cohort | Total
Number analyzed (Participants) | 23 | 9 | 32
Age, Continuous [Median (Full Range); unit: years] | 67 [36 to 82] | 70 [59 to 82] | 69 [36 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 18 | 7 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 23 | 8 | 31
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 20 | 8 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 9 | 32

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as at least a 20% increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) and the sum must also demonstrate an absolute increase of at least 5mm, or unequivocal progression of existing non-target lesions, or the appearance of new lesions. Estimated at 3 months using the Kaplan-Meier method.
Time Frame: 3 months
Population: Analysis population included those in the main Phase II study
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Afatinib)
Number analyzed (Participants) | 23
Participants | 5

2. Secondary Outcome: Overall Response Rate
Description: Includes both complete responses (CR) and partial responses (PR). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions: Complete Response (CR) is defined as the disappearance of all target lesions (any pathological lymph nodes must have reduction in short axis to <10 mm); Partial Response (PR) is defined as >=30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Overall Response (OR) = CR + PR.
Time Frame: Up to 3 years
Population: Analysis population includes those patients in the main Phase II study
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Afatinib)
Number analyzed (Participants) | 23
Participants | 2

3. Secondary Outcome: Median Progression-free Survival (PFS ) Time
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as at least a 20% increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) and the sum must also demonstrate an absolute increase of at least 5mm, or unequivocal progression of existing non-target lesions, or the appearance of new lesions. Estimated using the Kaplan-Meier method.
Time Frame: Up to 3 years
Population: Analysis population includes patients from the main Phase II study
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Afatinib)
Number analyzed (Participants) | 23
months | 1.4 [1.3 to 2.7]

4. Secondary Outcome: Median Overall Survival (OS) Time
Description: Estimated using the Kaplan-Meier method.
Time Frame: Up to 3 years
Population: Analysis population includes those in the main Phase II study
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Afatinib)
Number analyzed (Participants) | 23
months | 5.3 [3.7 to 7.4]

5. Secondary Outcome: EGFR Expression Status
Description: These analyses were conducted using available archival formalin-fixed, paraffin-embedded sections from surgical specimens. Each sample was tested to determine whether there was EGFR amplification.
Time Frame: Baseline
Population: The analysis sample included those in the main Phase II study. Two patients did not have a sample to analyze.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Afatinib)
Number analyzed (Participants) | 21
Participants | 5

6. Secondary Outcome: HER2 Expression Status
Description: These analyses were conducted using available archival formalin-fixed, paraffin-embedded sections from surgical specimens. Each sample was tested to determine whether there was HER2 amplification.
Time Frame: Baseline
Population: Analysis population included those in the main Phase II study. Two patients did not have a sample to analyze
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Afatinib)
Number analyzed (Participants) | 21
Participants | 4

7. Other Pre Specified Outcome: Presence of Tumor Micro Ribonucleic Acids (RNAs) Like miR-200
Description: Relationship to 3-month PFS will be determined.
Time Frame: Baseline
Population: This outcome measure was not assessed.
Arm/Group | Treatment (Afatinib)
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Epithelial to Mesenchymal Transition States
Time Frame: Up to 3 years
Population: This outcome measure was not assessed.
Arm/Group | Treatment (Afatinib)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the initiation of treatment to 28 days after the last administration of trial drugs, up to 1 year
Description: For the Other Adverse Events, the number of participants reported for each adverse event is an upper bound estimate.
Arm/Group | Treatment (Afatinib) - Phase II Study | Treatment (Afatinib) - Molecularly Selected Cohort
All-Cause Mortality (participants affected / at risk) | 21/23 | 9/9
Serious Adverse Events (participants affected / at risk) | 11/23 | 3/9
Other Adverse Events (participants affected / at risk) | 23/23 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Afatinib) - Phase II Study (N=23) | Treatment (Afatinib) - Molecularly Selected Cohort (N=9)
Small bowel obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Edema limbs (General disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
intracranial hemorrhage due to fall (Nervous system disorders) | 1 | 0
Skull fracture due to fall (Injury, poisoning and procedural complications) | 1 | 0
Altered mental status (Psychiatric disorders) | 1 | 0
Coughing up blood (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stent revision (Surgical and medical procedures) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Mouth sores (General disorders) | 0 | 1
Indiana pouch obstruction (Product Issues) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Afatinib) - Phase II Study (N=23) | Treatment (Afatinib) - Molecularly Selected Cohort (N=9)
Depression (Psychiatric disorders) | 4 | 1
Hypotension (Vascular disorders) | 2 | 1
Chronic kidney disease (Renal and urinary disorders) | 23 | 1
Proteinuria (Renal and urinary disorders) | 2 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 23 | 1
Dysgeusia (Nervous system disorders) | 3 | 1
Weight loss (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
Lipase increased (Investigations) | 0 | 1
INR increased (Investigations) | 6 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 1
Anemia (Blood and lymphatic system disorders) | 21 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Dizziness (General disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 1
Oral pain (Gastrointestinal disorders) | 1 | 1
General disorders - Other, specify (General disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 1
Mucositis oral (Gastrointestinal disorders) | 14 | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 3
Anorexia (Metabolism and nutrition disorders) | 22 | 5
Constipation (Gastrointestinal disorders) | 4 | 2
Diarrhea (Gastrointestinal disorders) | 23 | 9
Nausea (Gastrointestinal disorders) | 12 | 3
Vomiting (Gastrointestinal disorders) | 9 | 4
Fatigue (General disorders) | 23 | 8
Pain (General disorders) | 13 | 2
Alkaline phosphatase increased (Investigations) | 4 | 2
Creatinine increased (Investigations) | 10 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 3
Hyponatremia (Metabolism and nutrition disorders) | 3 | 3
Leukocytosis (Blood and lymphatic system disorders) | 6 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0
Ileal obstruction (Gastrointestinal disorders) | 3 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Fever (General disorders) | 5 | 0
Edema limbs (General disorders) | 6 | 0
Fracture (Injury, poisoning and procedural complications) | 2 | 0
Catheter related infection (Infections and infestations) | 2 | 0
Penile infection (Infections and infestations) | 5 | 0
Urinary tract infection (Infections and infestations) | 6 | 0
Confusion (Psychiatric disorders) | 4 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Intracranial hemorrhage (Nervous system disorders) | 2 | 0
Penile pain (Reproductive system and breast disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Urinary urgency (Renal and urinary disorders) | 2 | 0
Urinary tract pain (Renal and urinary disorders) | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 2 | 0
Hematuria (Renal and urinary disorders) | 11 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 0
Blood bilirubin increased (Investigations) | 3 | 0
Ejection fraction decreased (Investigations) | 4 | 0
Platelet count decreased (Investigations) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT02122172/Prot_SAP_000.pdf